CLINICAL TRIAL: NCT05004233
Title: Transmission Electron Microscopy Images for Platelet Ultrastructural Criteria Before and After the Onset of an Antiplatelet Agent
Acronym: ELECTROSTROKE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20CH026; 2021-A00292-39 (Other: ANSM)
Record Dates: First submitted 2021-07-16; First posted 2021-08-13 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke
Keywords: Ischemic stroke; Ultrastructural characterization; Transmission electron microscopy; platelet dysfunction; Blood Coagulation Disorder
MeSH Terms: conditions — Ischemic Stroke; Blood Coagulation Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ischemic stroke patients (Experimental): Patients hospitalized for an ischemic stroke.
  Interventions: Biological: Blood collection before antiplatelet treatment; Biological: Blood collection after antiplatelet treatment

INTERVENTIONS:
Biological: Blood collection before antiplatelet treatment — Blood sample (17ml) will be collected in the neurovascular department to be processed for platelet ultrastructural analysis before the onset of an antiplatelet treatment
Biological: Blood collection after antiplatelet treatment — A follow-up will be carried out 5 to 8 days after the initiation of the treatment.
  A blood test will be taken in the NeuroVascular Unit

SUMMARY:
The aim of the pilot study is to collect all the ultrastructural platelet characteristics by transmission electron microscopy before and after the onset of an antiplatelet treatment in patients hospitalized for an ischemic stroke ; and to assess recurrence of Ischemic Cerebral Accident (ICA) at 6 months in patients hospitalized for Ischemic stroke.

DETAILED DESCRIPTION:
Ischaemic stroke is the leading cause of adult disability. Thus, a strategy based on an efficient antiplatelet therapy has been developed to prevent platelet activation occurring in the acute phase of non-cardioembolic ischemic stroke.

The biological monitoring of the antiplatelet therapy with available platelet function assays do not provide a global integrative approach considering all the mechanisms involved in platelet activation.

Platelet transmission electron microscopy recently validated for assessing distinct ultrastructural abnormalities is a reliable morphological platelet structural analysis tool.

Ultrastructural criteria could be identified and be useful for the assessment of the degree of platelet activation and thus the biological efficiency of antiplatelet agents. All the activation transduction signals are integrated and all antiplatelet agents can be assessed.

The aim of the pilot study is to collect all the ultrastructural platelet characteristics by transmission electron microscopy before and after the onset of an antiplatelet treatment in patients hospitalized for an ischemic stroke.

Investigators expect to identify ultrastructural characteristics that will be correlated with the platelet degree of activation to guide clinicians in decision-making regarding the antiplatelet therapy strategy.

ELIGIBILITY:
Inclusion Criteria:

* Social security affiliation
* Signed informed consent
* patients hospitalized for an non cardioembolic ischemic stroke requiring the onset of an antiplatelet therapy according to the usual guidelines recommendations

Exclusion Criteria:

Contraindications regarding antiplatelet agent(s) and/or at least one excipient according to Summary of Product Characteristics (SPC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Morphology of the platelet : | Day 5
  Platelet ultrastructural criteria will be obtained from transmission electron microscopy images of platelet ultrathin sections before and after (5 days) initiation of antiaggregant therapy in patients with noncardioembolic ICA
  the morphology of the platelet :
  * discoid or round
  * with the emission of filipodia, pseudopodia and lamellipodia
Type of granules in the platelet | Day 5
  Platelet ultrastructural criteria will be obtained from transmission electron microscopy images of platelet ultrathin sections before and after (5 days) initiation of antiaggregant therapy in patients with noncardioembolic ICA
  - the observation of granules :
  * alpha granules
  * dense granules
Distribution of mitochondria, glycogen and dense tubular system in platelets | Day 5
  Platelet ultrastructural criteria will be obtained from transmission electron microscopy images of platelet ultrathin sections before and after (5 days) initiation of antiaggregant therapy in patients with noncardioembolic ICA
Structure of open canalicular system in platelets | Day 5
  Platelet ultrastructural criteria will be obtained from transmission electron microscopy images of platelet ultrathin sections before and after (5 days) initiation of antiaggregant therapy in patients with noncardioembolic ICA
  - the open canalicular system
  * dilated or not
  * associated with degranulation or not
Number of patients with a microtubular ring on the equatorial section plane (peripheral or centralized) in platelets | Day 5
  Platelet ultrastructural criteria will be obtained from transmission electron microscopy images of platelet ultrathin sections before and after (5 days) initiation of antiaggregant therapy in patients with noncardioembolic ICA

SECONDARY OUTCOMES:
The incidence of a composite endpoint | Month 6
  The incidence of a composite of cardiovascular events (radiologically documented recurrent ischemic stroke, transient ischemic attacks, coronary artery disease (acute coronary syndromes, myocardial infarction), obliterating arterial disease of the lower limb, death of cardiovascular origin)

CONTACTS AND LOCATIONS:
Overall Officials: PIERRE GARNIER, MD, Principal Investigator — CHU DE SAINT-ETIENNE
Locations (1):
- Centre Hospitalier Universitaire de St-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mallouk N, Garcin A, Li G, Epinat M, Szczepaniak C, Hien OF, Mismetti P, Garnier P. Platelet transmission electron microscopy for the assessment of poor biological response to antiplatelet agent: pilot descriptive and prospective study - ELECTROSTROKE. BMJ Open. 2022 Apr 4;12(4):e050060. doi: 10.1136/bmjopen-2021-050060. PMID 35379612